CLINICAL TRIAL: NCT07005687
Title: Using MSCs for Chronic Active Antibody Mediated Rejection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, nooshin dalili, MD, Shahid Beheshti University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBMU-1403
Record Dates: First submitted 2024-05-29; First posted 2025-06-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Kidney Transplant Rejection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSCs Derived (Other)
  Interventions: Other: Stem Cells

INTERVENTIONS:
Other: Stem Cells — MSCs Derived

SUMMARY:
Mesenchymal stem cell (MSCs) therapy has already been studied in kidney transplant recipients (KTRs), and the available data showed that it is safe and well tolerated. The aim of this study was to evaluate the safety and efficacy of autologous MSCs in combination with standard therapy in KTRs with biopsy-proven chronic active antibody-mediated rejection (AMR). Patients with biopsy-proven chronic active AMR received treatment with autologous bone marrow-derived MSCs (3 × 106 cells/kg iv) after completion of standard therapy and were followed for up to 12 months. The primary endpoints were safety by assessment of adverse events. Secondary endpoints included assessment of kidney graft function, immunological and histological changes related to AMR activity and chronicity assessed by conventional microscopy and molecular transcripts. A total of 3 patients were enrolled in the study before it was terminated prematurely because of adverse events. We found that AMR did not improve in any of the patients after treatment with MSCs. In addition, serious adverse events were observed in one case when autologous MSCs therapy was administered in the late phase after kidney transplantation, which requires further elucidation.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the safety and efficacy of autologous MSCs in combination with standard therapy in KTRs with biopsy-proven chronic active antibody-mediated rejection (AMR). Patients with biopsy-proven chronic active AMR will receive treatment with autologous bone marrow-derived MSCs (3 × 106 cells/kg iv) after completion of standard therapy and will be followed for up to 12 months. The primary endpoints are safety by adverse events. Secondary endpoints include assessment of kidney graft function, immunological and histological changes related to AMR activity and chronicity assessed by conventional microscopy and molecular transcripts.

ELIGIBILITY:
Inclusion Criteria:

* chronic active antibody mediated rejection in kidney transplanted recipients

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2027-12-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
progression of chronicity index | one year after administration
  Number of participants with treatment-related adverse events as assessed by kidney biopsy

IPD SHARING:
Plan to Share IPD: No